CLINICAL TRIAL: NCT01655901
Title: Effects of Active Video Games on Energy Balance: a Randomized Crossover Study in Adolescents
Brief Title: Active Video Games and Appetite Control in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jean-Philippe Chaput, Junior Research Chair, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 272112
Record Dates: First submitted 2012-07-30; First posted 2012-08-02 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Active Video Games and Appetite Control
Keywords: Active video games; Food intake; Energy balance; Adolescents
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active video gaming (Experimental): Playing Kinect
  Interventions: Behavioral: Active video gaming; Behavioral: Passive video gaming; Behavioral: Resting
- Passive video gaming (Experimental): Playing Xbox 360
  Interventions: Behavioral: Active video gaming; Behavioral: Passive video gaming; Behavioral: Resting
- Resting (Experimental): Stay seated on a comfortable chair
  Interventions: Behavioral: Active video gaming; Behavioral: Passive video gaming; Behavioral: Resting

INTERVENTIONS:
Behavioral: Active video gaming
Behavioral: Passive video gaming
Behavioral: Resting

SUMMARY:
STATEMENT OF THE PROBLEM: Video games have enormous mass appeal, are omnipresent in the daily schedule of most children and youth and have been linked to the obesity epidemic. The investigators research group recently reported that sedentary video game playing increases food intake in adolescents. Interestingly, the overconsumption of food associated with seated video game play was observed without increased sensations of hunger and appetite, as previously observed with television viewing. Active video games offer an appealing opportunity for increasing energy expenditure and promoting healthy body weight among children and youth who might otherwise be spending time in sedentary screen-based activities. However, significant increases in energy expenditure as a result of active video game play might be of little importance to energy balance if one compensates by increasing energy intake and/or decreasing physical activity. Studies to date have failed to measure energy intake so it is currently unknown the effects of active video games on daily energy balance.

OBJECTIVE: The main aim of this study is to examine the acute effects of playing active video games on energy intake and expenditure.

HYPOTHESIS: The investigators hypothesize that the increase in energy expenditure promoted by active video games will be offset by compensatory adjustments in food intake and spontaneous physical activity subsequent to the intervention.

RESEARCH PLAN: With the use of a randomized crossover design, 30 normal-weight and 30 obese adolescents between 13 and 17 years of age will complete three 1-hour experimental conditions, namely (1) resting in a sitting position (control condition), (2) playing Xbox 360 (sedentary video game condition) and (3) playing Kinect (active video game condition), followed by an ad libitum lunch. The primary outcomes will be acute (24-h) and short-term (3-day) energy intake and expenditure. Food intake will be measured using an ad libitum test meal immediately following the intervention, a food menu for the remainder of the day and a dietary record for the subsequent 3-day period. Energy expenditure will be measured using indirect calorimetry during the intervention and an Actical accelerometer for the subsequent 3-day period. Secondary outcomes will include appetite sensations (visual analogue scales), stress markers (heart rate variability, blood pressure, and mental workload), and levels of appetite-related hormones and substrates (glucose, insulin, cortisol, leptin, and ghrelin).

RELEVANCE: The present study is innovative and likely to result in a number of new and important findings that can inform future recommendations. If the investigators confirm our hypothesis, the clinical implication will be to rethink the strategy of promoting active video games as an intervention tool for the prevention of overweight and obesity in youth.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between the ages of 13 and 17

Exclusion Criteria:

* Current smoker
* Unstable body weight (±4 kg) during the 6 months preceding testing
* Excessive intake of alcohol (>10 drinks/week) or substance abuse
* Metabolic disease (e.g. thyroid disease, heart disease, diabetes, etc)
* Celiac disease or vegetarian
* Medication use that could interfere with the outcome variables
* Highly restrained eating behavior
* Irregular eating pattern (e.g. skipping breakfast)
* Unfamiliar with the use of video games
* Inability to comply with the protocol

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Chaput, PhD, Principal Investigator — Children's Hospital of Eastern Ontario Research Institute
Locations (1):
- Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Chaput JP, Visby T, Nyby S, Klingenberg L, Gregersen NT, Tremblay A, Astrup A, Sjodin A. Video game playing increases food intake in adolescents: a randomized crossover study. Am J Clin Nutr. 2011 Jun;93(6):1196-203. doi: 10.3945/ajcn.110.008680. Epub 2011 Apr 13. PMID 21490141
- [Derived] Gribbon A, McNeil J, Jay O, Tremblay MS, Chaput JP. Active video games and energy balance in male adolescents: a randomized crossover trial. Am J Clin Nutr. 2015 Jun;101(6):1126-34. doi: 10.3945/ajcn.114.105528. Epub 2015 Mar 11. PMID 25762809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized crossover study (1 group doing all 3 conditions). Wash-out period of 1 week between conditions.
Groups:
- Kinect, Then Xbox360, Then Sitting: Participants played Kinect for 1 hour at 10:20am. After a wash-out period of 1 week, they then played Xbox360 for 1 hour at 10:20am. After a second wash-out period of 1 week they then sat on a chair for 1 hour at 10:20am.
- Kinect, Then Sitting, Then Xbox360: Participants played Kinect for 1 hour at 10:20am. After a wash-out period of 1 week, they then sat on a chair for 1 hour at 10:20am. After a second wash-out period of 1 week they then played Xbox360 for 1 hour at 10:20am.
- Xbox360, Then Sitting, Then Kinect: Participants played Xbox360 for 1 hour at 10:20am. After a wash-out period of 1 week, they then sat on a chair for 1 hour at 10:20am. After a second wash-out period of 1 week they then played Kinect for 1 hour at 10:20am.
- Xbox360, Then Kinect, Then Sitting: Participants played Xbox360 for 1 hour at 10:20am. After a wash-out period of 1 week, they then played Kinect for 1 hour at 10:20am. After a second wash-out period of 1 week they then sat on a chair for 1 hour at 10:20am.
- Sitting, Then Kinect, Then Xbox360: Participants sat on a chair for 1 hour at 10:20am. After a wash-out period of 1 week, they then played Kinect for 1 hour at 10:20am. After a second wash-out period of 1 week they then played Xbox360 for 1 hour at 10:20am.
- Sitting, Then Xbox360, Then Kinect: Participants sat on a chair for 1 hour at 10:20am. After a wash-out period of 1 week, they then played Xbox360 for 1 hour at 10:20am. After a second wash-out period of 1 week they then played Kinect for 1 hour at 10:20am.
Period: First Intervention (Hour 1)
Arm/Group | Kinect, Then Xbox360, Then Sitting | Kinect, Then Sitting, Then Xbox360 | Xbox360, Then Sitting, Then Kinect | Xbox360, Then Kinect, Then Sitting | Sitting, Then Kinect, Then Xbox360 | Sitting, Then Xbox360, Then Kinect
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Kinect, Then Xbox360, Then Sitting | Kinect, Then Sitting, Then Xbox360 | Xbox360, Then Sitting, Then Kinect | Xbox360, Then Kinect, Then Sitting | Sitting, Then Kinect, Then Xbox360 | Sitting, Then Xbox360, Then Kinect
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Hour 2)
Arm/Group | Kinect, Then Xbox360, Then Sitting | Kinect, Then Sitting, Then Xbox360 | Xbox360, Then Sitting, Then Kinect | Xbox360, Then Kinect, Then Sitting | Sitting, Then Kinect, Then Xbox360 | Sitting, Then Xbox360, Then Kinect
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Kinect, Then Xbox360, Then Sitting | Kinect, Then Sitting, Then Xbox360 | Xbox360, Then Sitting, Then Kinect | Xbox360, Then Kinect, Then Sitting | Sitting, Then Kinect, Then Xbox360 | Sitting, Then Xbox360, Then Kinect
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (Hour 3)
Arm/Group | Kinect, Then Xbox360, Then Sitting | Kinect, Then Sitting, Then Xbox360 | Xbox360, Then Sitting, Then Kinect | Xbox360, Then Kinect, Then Sitting | Sitting, Then Kinect, Then Xbox360 | Sitting, Then Xbox360, Then Kinect
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 4 | 4 | 5 | 4 | 5
Not Completed | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Completers analyzed
Groups:
- Video Game Condition: Playing Kinect
  Playing Xbox 360
  Sitting on a chair (control)
Arm/Group | Video Game Condition
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 26
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 21.8 (5.0)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] | 74.1 (12.7)
Resting metabolic rate (kJ/day) [Mean (Standard Deviation); unit: kJ/day] | 7101 (1224)
Tanner puberty stages (self-assessed by questionnaire) [Mean (Standard Deviation); unit: units on a scale] — Self-assessment questionnaire that aims to measure pubertal status by using line drawings of the Tanner puberty stages. Scores range from 1 to 5 for genitals and pubic hair development (5 being more developed).
  units on a scale | 3.5 (0.9)
Physical Activity Questionnaire score [Mean (Standard Deviation); unit: units on a scale] — The Physical Activity Questionnaire for Adolescents, a self-report measure of physical activity, was used to assess physical activity level. A score of 1 and a score of 5 indicate low and high physical activity participation, respectively.
  units on a scale | 2.3 (0.5)
Cohen's Perceived Stress Scale score [Mean (Standard Deviation); unit: units on a scale] — The Cohen's Perceived Stress Scale was completed to evaluate the amount of stress in the participant's daily life. This questionnaire contains 10 questions and a score of less than 10 indicates good stress management. The scale goes from 0 to 40, with higher scale scores indicating poor stress management.
  units on a scale | 13.0 (5.4)
Pittsburgh Sleep Quality Index score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index was completed by participants. This self-rated questionnaire assesses sleep quality and disturbances over the preceding month. It contains 21 questions and a score greater than 5 is associated with poor sleep. The scores range from 0 to 21, with higher scores indicating poor sleep quality.
  units on a scale | 4.8 (2.3)
Levels of appetite-related hormones [Mean (Standard Deviation); unit: mmol/L] — Profiles of glucose, insulin, cortisol, leptin, and ghrelin. Even this assessment was originally planned no measures were finally taken due to financial constraints. Because the data were not collected no data could be reported. Population: Data were not collected

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake and Energy Expenditure (Over 24 Hours and Over 3 Days)
Description: Energy intake (kJ) was measured using an ad libitum test meal immediately following the 3 experimental conditions, a food menu for the remainder of the day, and a dietary record for the subsequent 3-day period. Energy expenditure was measured by indirect calorimetry during the 3 experimental conditions, and by using an Actical accelerometer for the subsequent 3-day period.
Time Frame: Acute (24 hours) and short-term (3 days)
Measure: Mean (Standard Error); unit: kJ
Groups:
- All Study Participants: Active video gaming (Kinect) Passive video gaming (Xbox360) Sitting on a chair (control)
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
kJ
  Energy intake Kinect 24 hours | 17981 (10104)
  Energy intake Xbox360 24 hours | 17014 (10023)
  Energy intake control 24 hours | 17566 (9984)
  Energy expenditure Kinect 24 hours | 10413 (567)
  Energy expenditure Xbox360 24 hours | 9581 (562)
  Energy expenditure control 24 hours | 9598 (558)
  Energy intake Kinect 3 days | 31412 (4123)
  Energy intake Xbox360 3 days | 35412 (3967)
  Energy intake control 3 days | 3346 (4043)
  Energy expenditure Kinect 3 days | 30997 (1456)
  Energy expenditure Xbox360 3 days | 30498 (1489)
  Energy expenditure control 3 days | 30141 (1534)

2. Secondary Outcome: Appetite Sensation
Description: Visual analogue scale to assess appetite feelings. The scale is 100 mm in length and ranges from 0 mm (not hungry at all) to 100 mm (extremely hungry).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mm
Groups:
- All Study Participants: Active video gaming (Kinect)
  Passive video gaming (Xbox360)
  Resting (control)
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
mm
  Kinect | 51 (53)
  Xbox360 | 56 (54)
  Control | 58 (49)

3. Secondary Outcome: Stress Marker
Description: Mental effort assessed on a visual analogue scale (100 mm in length). It ranges from 0 mm (no mental effort at all) to 100 mm (extremely mentally challenging).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mm
Groups:
- All Study Participants: Active video gaming (Kinect)
  Passive video gaming (Xbox)
  Resting (control)
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
mm
  Kinect | 52 (45)
  Xbox360 | 54 (56)
  Control | 43 (42)

4. Secondary Outcome: Levels of Appetite-related Hormones
Description: Profiles of glucose, insulin, cortisol, leptin, and ghrelin assessed at every 10 minutes during each 1-hour experimental condition.
Time Frame: 1 hour
Population: Not analyzed due to lack of funds (major budget cut)
Groups:
- All Study Participants: Active video gaming (Kinect)
  Passive video gaming (Xbox 360)
  Resting (control)
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Kinect: Participants played Kinect for 1 hour at 10:20am.
- Xbox360: Participants played Xbox360 for 1 hour at 10:20am.
- Sitting: Participants sat for 1 hour at 10:20am.
Arm/Group | Kinect | Xbox360 | Sitting
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No